CLINICAL TRIAL: NCT00893217
Title: Double-blind, Randomized, Parallel Group, Multicenter Study of the Safety and Tolerability of Betaseron 500 Mcg Subcutaneously Every Other Day and Betaseron 250 Mcg Subcutaneously Every Other Day for at Least 12 Weeks in Patients With RRMS
Brief Title: BEYOND Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Healthcare Pharmaceuticals Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91232; BEYOND pilot; 307000
Record Dates: First submitted 2009-05-04; First posted 2009-05-05 (Estimated); Last update posted 2009-11-09 (Estimated); Status verified 2009-11

CONDITIONS: Multiple Sclerosis; Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: Betaseron (Interferon beta-1b, BAY86-5046)
- Arm 2 (Experimental)
  Interventions: Drug: Betaseron (Interferon beta-1b, BAY86-5046)

INTERVENTIONS:
Drug: Betaseron (Interferon beta-1b, BAY86-5046) — 250 mcg
  Arms: Arm 1
Drug: Betaseron (Interferon beta-1b, BAY86-5046) — 500 mcg
  Arms: Arm 2

SUMMARY:
The purpose of this study is to valuate safety and tolerability of Betaseron.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of RRMS as defined by any of the following McDonald diagnostic criteria (McDonald et al 2001; see Appendix 16.1.1 [(Protocol Appendix 5]):

* Two relapses and objective clinical evidence (history or present) of at least 2 lesions
* Two relapses and objective clinical evidence (history or present) of 1 lesion; and dissemination in space, demonstrated by MRI (Barkhof/Tintoré criteria) or 2 MRI T2 lesions consistent with MS plus positive CSF.
* One relapse with objective clinical evidence (history or present) of at least 2 lesions, and dissemination in time, demonstrated signs of disease activity ( new Gd+ lesion or new T2 lesion) in an MRI scan at least 3 months after the onset of that clinical event.
* One relapse and objective clinical evidence (history or present) of 1 lesion, and dissemination in space, demonstrated by MRI (Barkhof/Tintoré criteria); or 2 MRI T2 lesions consistent with MS plus positive CSF, and dissemination in time, demonstrated by signs of disease activity (new Gd+ lesion or new T2 lesion) in an MRI scan at least 3 months after the onset of that clinical event.

  * 18 to 55 years of age
  * Score of 0-5.5 on the Kurtzke Expanded Disability Status Scale' (EDSS; see Appendix 16.1.1 [Protocol Appendix 4])
  * Naïve to immunomodulating therapies or previously treated with immunomodulating therapies other than any interferon (IFN) more than 30 days prior to the start of the study
  * If female of child-bearing potential, agreement to practice adequate contraception methods (IUCD, condoms, oral contraceptives, or other adequate barrier contraception)
  * Negative serum pregnancy test results.
  * Signed and dated statement of informed consent

Exclusion Criteria:

* Clinically significant heart disease such as uncontrolled cardiac dysrhythmia, angina pectoris, cardiomyopathy, or congestive heart failure
* History of severe depression, suicide attempts, or current suicidal ideations
* Clinically significant liver, renal, and bone marrow dysfunction as defined by any of the following laboratory evaluations:
* bone marrow dysfunction:

  * Hb <8.5 g/dl
  * WBC <2.5 x 109/L
  * platelet count <125 x 109/L
* renal dysfunction: creatinine >1.8 mg/dL
* liver dysfunction:

  * ASAT (SGOT) >3xupper limit of normal
  * bilirubin >2x upper limit of normal
* Epilepsy not adequately controlled by treatment
* Any conditions that could interfere with the MRI or any other evaluation in the study
* Known allergy to human proteins including albumin and IFN, or to mannitol or gadolinium
* Participation in any clinical study within the past 30 days or use/intake of an investigational drug within the last 3 months prior to study entry
* Prior treatment with monoclonal antibody therapy, cladribine or total lymphoid irradiation
* Treatment with cytotoxic or immunosuppressive therapies (except systemic steroid or adrenocorticotropic hormone [ACTH]) within 6 months prior to study entry; or systemic steroid or ACTH within 1 month prior to study entry
* Presence of monoclonal gammopathy
* Inability to tolerate both NSAIDs and acetaminophen
* Pregnancy or lactation
* History of alcohol or drug abuse
* Inability to administer subcutaneous injections either by self or by caregiver
* Medical, psychiatric or other conditions that compromise the patient's ability to give informed consent, to understand the patient information, to comply with the study protocol, or to complete the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2002-11; Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of IFNB-1b 500 mcg given subcutaneously (SC) QOD compared with the standard dose of 250 mcg QOD in patients with RRMS. | 8 Months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (14):
- United States (14):
  - Los Angeles, California
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - Chicago, Illinois
  - Kansas City, Kansas
  - Louisville, Kentucky
  - Ann Arbor, Michigan
  - Reno, Nevada
  - Stony Brook, New York
  - Durham, North Carolina
  - High Point, North Carolina
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Nashville, Tennessee